CLINICAL TRIAL: NCT06974643
Title: Thoracic Epidural Anesthesia Versus Paravertebral Block for Awake Thoracotomy: A Randomized Non-inferiority Trial
Brief Title: Thoracic Epidural Anesthesia Versus Paravertebral Block for Awake Thoracotomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Elsaid Abdel Fattah, Lecturer of Anesthesia, Surgical ICU and Pain Management, Faculty of Medicine, National Cancer Institute, Cairo University, Egypt., Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AP2503-501-099-197
Record Dates: First submitted 2025-05-08; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Thoracic Epidural Anesthesia; Paravertebral Block; Awake Thoracotomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thoracic epidural block group (Experimental): Patients will preoperatively receive an awake thoracic epidural block.
  Interventions: Other: Thoracic epidural block
- Paravertebral block group (Experimental): Patients will preoperatively receive a paravertebral block.
  Interventions: Other: Paravertebral block

INTERVENTIONS:
Other: Thoracic epidural block — Patients will preoperatively receive an awake thoracic epidural block.
  Arms: Thoracic epidural block group
Other: Paravertebral block — Patients will preoperatively receive a paravertebral block.
  Arms: Paravertebral block group

SUMMARY:
This study aims to compare paravertebral block and thoracic epidural in awake thoracotomy.

DETAILED DESCRIPTION:
Pain can often persist after thoracotomy, and the incidence of chronic pain is high, with studies revealing that 30% to 50% of patients still experience pain up to five years after surgery.

Thoracic epidural blockade (TEB) blocks nerves that supply the chest with local anesthetic bilaterally, at the spinal cord level. It acts by reducing the onward transmission of painful nerve signals, but may not abolish them altogether. Paravertebral blockade (PVB) involves injecting local anesthetic into the paravertebral space, which contains spinal nerves (and sometimes even extension of the dura), white and grey rami communicantes, the sympathetic chain, and intercostal vessels, on the side of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 60 years.
* Both genders.
* American Society of Anesthesiologists (ASA) physical status classification II or III.
* Scheduled for thoracotomy.

Exclusion Criteria:

* Poor cardiac function (ejection fraction less than 50%).
* Patients with bad pulmonary function testing (PFTs). Absolute contraindication to thoracic epidural anesthesia includes patient refusal, allergy to local anesthetics, coagulopathy, active neurologic disorders, skin infection at the insertion site, uncooperative patients, uncontrolled cough, and unfavorable anatomy for thoracic epidural.
* Thoracic spine disorders require chest wall resection or emergency thoracic surgery.
* Had a previous thoracotomy (scarring due to prior surgery can limit the effectiveness of paravertebral block, and these patients may have existing chronic pain).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Intraoperative fentanyl consumption | Intraoperatively
  Additional bolus doses of fentanyl 0.5µg/kg will be given if the mean arterial blood pressure or heart rate rises above 20% of baseline levels.

SECONDARY OUTCOMES:
Time to the 1st rescue analgesia | 48 hours postoperatively
  Time to first request of rescue analgesia will be assessed from the end of surgery till first dose of morphine administrated.
Mean arterial pressure | Till the end of surgery (Up to 2 hours)
  Mean arterial pressure will be recorded at baseline, and every 15min till the end of surgery
Heart rate | Till the end of surgery (Up to 2 hours)
  Heart rate will be recorded at baseline, and every 15min till the end of surgery
Total morphine consumption | 48 hours postoperatively
  If numeric rating scale (NRS)>3 at rest will be observed, rescue analgesia via IV morphine 3 mg boluses will be administered.
Degree of pain | 48 hours postoperatively
  The patients will be instructed how to report pain by the numeric rating scale (NRS) [on a scale from (0 to 10), zero means no pain and ten means the worst pain]. NRS will be measured at post-anesthesia care unit (PACU), 1, 2, 4, 8, 12, 18, 24, 36, 48 hours postoperatively at rest and movement
Degree of patient satisfaction | 48 hours postoperatively
  Degree of patient satisfaction will be assessed on a 5-point Likert scale patient satisfaction (1, extremely dissatisfied; 2, unsatisfied; 3, neutral; 4, satisfied; 5, extremely satisfied)
Incidence of adverse events | 48 hours postoperatively
  Incidence of adverse events such as nausea, vomiting, respiratory depression, hypotension and bradycardia

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.